CLINICAL TRIAL: NCT06020235
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Study to Evaluate Safety and Antimicrobial Efficacy of Topically Once or Twice Daily Applied Bisphosphocin® Nu-3 Gel At 5% and 10% Concentrations to Infected Diabetic Foot Ulcers (iDFU)
Brief Title: Nu-3 Gel for Infected Diabetic Foot Ulcers
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lakewood-Amedex Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAI-Nu-3-CLIN004
Record Dates: First submitted 2023-08-08; First posted 2023-08-31 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Foot Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 5% Nu-3 gel once daily (Experimental): The 5% Nu-3 gel is applied once per day and placebo is applied once per day.
  Interventions: Drug: 5% Nu-3 gel; Drug: Placebo
- 5% Nu-3 gel twice daily (Experimental): The 5% Nu-3 gel is applied twice per day.
  Interventions: Drug: 5% Nu-3 gel
- 10% Nu-3 gel once daily (Experimental): The 10% Nu-3 gel is applied once per day and placebo is applied once per day.
  Interventions: Drug: 10% Nu-3 gel; Drug: Placebo
- 10% Nu-3 gel twice daily (Experimental): The 10% Nu-3 gel is applied twice per day.
  Interventions: Drug: 10% Nu-3 gel
- Placebo (Placebo Comparator): The placebo is applied twice per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5% Nu-3 gel — The gel is called Nu-3 which is either applied once per day or twice per day to the infected ulcer.
  Arms: 5% Nu-3 gel once daily; 5% Nu-3 gel twice daily
Drug: 10% Nu-3 gel — The gel is called Nu-3 which is either applied once per day or twice per day to the infected ulcer.
  Arms: 10% Nu-3 gel once daily; 10% Nu-3 gel twice daily
Drug: Placebo — Placebo gel is either applied once per day or twice per day to the infected ulcer.
  Arms: 10% Nu-3 gel once daily; 5% Nu-3 gel once daily; Placebo

SUMMARY:
The goal of this clinical trial is to test a topical drug in patients with mild infections of their diabetic foot ulcer. The main questions it aims to answer are:

What strength does the drug need to be in order to make the infection better? How frequently does the drug need to be applied in order to make the infection better? Participants will be asked to apply the medicine on their foot ulcer twice a day for 2 weeks and remain off of that foot during that time.

Participants will receive the medication either once a day or twice a day, in either a 5% or 10% gel, or placebo.

Researchers will compare the 5% and 10% gels to placebo to see if the infection improves.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male and female subjects ≥18 years of age. 2. Voluntary written informed consent, including information about the provisions of the Health Insurance Portability and accountability act (HIPAA) as applicable.

  3. Non-hospitalized ambulatory subjects diagnosed with diabetes mellitus, Type I or II per ADA criteria with signs of a localized mild foot infection as defined by the IDSA infection severity criteria (Lipsky,2012)

  a. the presence of purulent drainage or at least two of the following criteria: i. erythema, ii. warmth, iii. pain or tenderness, iv. edema, or v. induration (The diagnosis of mild infection must be confirmed immediately following debridement at Baseline).

  4. The target ulcer is classified as a grade 1 ulcer according to the Wagner Scale (Wagner 1979). The ulcer is a superficial, full-thickness ulcer limited to the dermis, not extending to the subcutis. Target ulcer is >1 cm2 and <12 cm2 post debridement at baseline and must be no higher than the ankle, on or below the malleolus (ankle bone) with ≥50% below the malleolus.

  5. Adequate vascular perfusion as evidenced by one of the following:
  1. Dorsal transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 40 mmHg
  2. Ankle Branchial Index (ABI) between 0.9 and 1.3 within 3 months of Screening using the extremity with the target ulcer.
  3. Arterial Doppler ultrasound evaluating for biphasic or triphasic dorsalis pedis and posterior tibial vessels at the level of the ankle or a TBI (Toe Brachial Index) of >0.75.

     6. Subject has a caregiver who will attend the Baseline visit (V2) and/or watch the dosing and dressing demonstration video and apply wound treatment along with study dressings for the study duration.

     7. Must meet one of the following criteria:

  a. Female subjects of Non-Child-Bearing Potential i. Postmenopausal for at least 1 year ii. Surgically sterilized (i.e., hysterectomy or bilateral oophorectomy more than 3 months prior to Screening) iii. Bilateral tube ligation > 6 months prior to screening iv. A negative serum β-hCG pregnancy test at screening and no breastfeeding after the administration of the study drug.

  b. Male subjects of Non-Childbearing Potential defined as: i. Vasectomized subjects for > 6 months prior to Screening ii. Those diagnosed as sterile by a physician. c. Females and Males of Childbearing Potential who practice an acceptable method of contraception defined as the i. Use of any form of hormonal contraceptive ii. Use of a barrier method with spermicide, condoms, intrauterine device, iii. Abstinence from sexual intercourse starting at least 60 days prior to Screening and continuing at least 14 days following the last treatment.

  8. Subjects must be willing to undergo all clinical investigation-related procedures, attend all required visits, and cooperate fully with the investigator and site personnel.

  9. Subject must be willing to wear offloading RCW, if necessary, throughout the duration of the clinical treatment.

  10. Subject must have plain radiograph taken at screening and prior to randomization showing no evidence of bony abnormalities consistent with osteomyelitis, or gas compatible with tissue crepitus, in the affected foot.

Exclusion Criteria:

* 1. Ulceration with exposed tendon, capsule, or bone 2. IDSA-defined moderate or severe DFU infection. 3. Infected diabetic foot ulcer that is associated with local wound complication such as prosthetic materials or protruding surgical hardware.

  4. > 1 infected foot ulcer 5. Subject is currently receiving topical antimicrobial treatment for a localized infection of the study ulcer and whose infection is improving in response to treatment.

  6. Subject has received a systemic antibiotic within 48 hours prior to Screening.

  7. Concurrent or expected to require systemic antimicrobials during the study period for any infection including diabetic foot ulcer.

  8. Any subject that has active viral hepatitis (A, B, C) and/or untreated HIV/AIDS.

  9. Any subject that has vascular compromise requiring surgical intervention or has undergone vascular reconstruction or angioplasty less than 1 month prior to randomization. Any planned surgical procedures during the study participation 10. eGFR <60 and/or subject on hemodialysis within 3 months prior to randomization.

  11. Hemoglobin A1c (HbA1c) >12% within 3 months prior to randomization. 12. Aspartate Aminotransferase (AST, GOT) and/or Alanine Aminotransferase (ALT, GPT) >3.0 x the upper limit of normal and/or bilirubin >1.5 x the upper limit of normal within 3 months prior to randomization.

  13. Acute active Charcot foot 14. Any subject that would be unable to safely monitor the infection status at home and return for scheduled visits.

  15. History of immunosuppression within 3 months prior to randomization, or taking immunosuppressive agents including systemic corticosteroids, except stable daily doses of 5 mg/day or less for chronic conditions 16. Any subject with a life expectancy ≤ 6 months 17. Use of investigational drugs within 28 days prior to screening 18. Use of Aspirin® or acetylsalicylic acid containing medication (except low-dose aspirin) < 7 days before baseline, 19. Use of oral anticoagulants (e.g., warfarin, Xarelto® or comparable products).

  20. History of concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol including known or suspected active abuse of alcohol, narcotics, or non-prescription drugs.

  21. Prior randomization in this clinical trial, or a previous Bisphosphocin study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Safety | Day 0 to Day 28
  Number of AEs overall and those assessed by the investigators as possibly, probably, and definitely related to the study drug; number of SAEs per patient and cohort
Efficacy | Day 0 to Day 14
  The rate of reduction in CFUs by >=2 logs per pathogen identified as typical and highly suspicious for being the cause of the infection, in each treatment group compared to placebo group at Day 7 compared to Day 0, and Day 14 compared to Day 0.

SECONDARY OUTCOMES:
Treatment failure rate per treatment regimen | Day 0 to Day 14
  The proportion of patients whose infection was not cured, defined as resolution of all wound infection signs, or whose infection did not improve over the course of the study defined as a lower number of clinical signs of infection or lower extent or severity as assesed by wound infection score.
Treatment failure rate per treatment regimen | Day 0 to Day 14
  Number of treatment failures, defined as need to switch to oral antibiotic treatment based on clinical wound-infection assessment by the PI, per cohort
Safety | Day 0 to Day 28
  Number of AEs (overall and those assessed by the investigators as possibly, probably and definitely related to the study drug) and SAEs per patient and cohort and clinically relevant changes in physical examination, vital signs, laboratory and/or ECG measurements at the defined timepoints compared to baseline
Safety | Day 0 to Day 28
  Change in parameters indicative of skin irritation and/or skin sensitization compared to baseline
Pharmacokinetics | Day 0 to Day 13
  Maximum concentration in the first 20 patients sampled for PK across all dosing groups after initial and repeated dosing

OTHER OUTCOMES:
Wound healing | Day 0 to Day 28
  Percentage area reduction of wound size at Day 7, Day 14, and Day 28 compared to baseline
Wound healing | Day 0 to Day 28
  Change in the 5-component clinical signs DFI score at all timepoints compared to baseline
Wound healing | Day 0 to Day 28
  Change in the overall DFI score at all timepoints compared to baseline

IPD SHARING:
Plan to Share IPD: No